CLINICAL TRIAL: NCT06925932
Title: Reducing Free Sugar Intakes - The Role of Sweet Taste III
Brief Title: This Trial Aims to Assess the Effects of Three Different Taste-based Dietary Recommendations for Reducing Free Sugar Intakes on Free Sugar Consumption in UK High Free Sugar Consumers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BielatRCT2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Dietary Behavior; Free Sugar; Sweet Taste
Keywords: dietary behavior; free sugar; sweet taste

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and all outcome assessors will be blinded to the intervention allocation. Participants will also be blinded to intervention allocation aside from their own. Data processing and analysis will be undertaken in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sweet taste arm (Active Comparator): Description: Participants in this arm will be asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are sweet but have no or low amounts of free sugars, e.g., sweet no- or low-free sugar foods, fruit, and no- or low-calorie sweeteners.
  Interventions: Behavioral: Dietary advice - Sweet taste
- Taste arm (Active Comparator): Description: Participants in this arm will be asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are non-sweet but are full of tasty flavours, e.g., non-sweet foods and drinks with nuts, herbs or spices.
  Interventions: Behavioral: Dietary advice - Taste
- No taste arm (Active Comparator): Description: Participants in this arm will be asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are non-sweet and have no strong flavours, e.g., non-sweet plain foods and drinks.
  Interventions: Behavioral: Dietary advice - No taste

INTERVENTIONS:
Behavioral: Dietary advice - Sweet taste — Asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are sweet but have no or low amounts of free sugars, e.g., sweet no- or low-free sugar foods, fruit, and no- or low-calorie sweeteners.
  Arms: Sweet taste arm
Behavioral: Dietary advice - Taste — Asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are non-sweet but are full of tasty flavours, e.g., non-sweet foods and drinks with nuts, herbs or spices.
  Arms: Taste arm
Behavioral: Dietary advice - No taste — Asked to reduce their free sugar intakes to < 5%TEI and replace sweet foods and drinks that are high in free sugars with foods and drinks that are non-sweet and have no strong flavours, e.g., non-sweet plain foods and drinks.
  Arms: No taste arm

SUMMARY:
This randomised controlled trial aims to assess the effects of three different taste-based dietary recommendations for reducing free sugar intakes on free sugar consumption in UK high free sugar consumers.

DETAILED DESCRIPTION:
This 12-week, 3-arm randomised controlled trial aims to assess the effects of three different taste-based food and beverage substitution instructions for reducing free sugar intakes on free sugar consumption in high free sugar consumers. A total of 180 adult community members residing in Bournemouth and the surrounding areas will be recruited. All participants will be asked to reduce their intakes of free sugar and replace sweet, high-free sugar foods and beverages with either: 1) sweet tasting foods and beverages that have no or low amounts of free sugars; 2) non-sweet tasting foods and beverages that have no or low amounts of free sugars and are high in other tasty flavours; and 3) non-sweet tasting foods and beverages that have no or low amounts of free sugars and are also low in other flavours. The primary outcome of interest is the changes in free sugar intakes from baseline to endpoint. Secondary outcomes include a range of dietary and biopsychosocial outcomes, sweet taste perceptions and sweet food and beverage intakes, as well as compliance with and evaluation of the dietary recommendation received.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over
2. Consuming more than 10% total daily energy from free sugars (-3% for testing error)
3. Residing in the South of England, and able to attend Bournemouth University for testing (Talbot Campus, BH12 5BB)
4. Able to provide consent and complete all study-related measures

Exclusion Criteria:

1. Being a smoker or having smoked in the last 3 months
2. Being pregnant or breastfeeding
3. Being underweight (BMI < 18.5 kg/m²)
4. Dieting or following a specific diet program (e.g., Weight Watchers, Keto diet, or Intermittent Fasting)
5. Following a specific diet or nutritional advice as a result of pre-existing medical condition (e.g., Crohn's disease, diabetes)
6. Having a pre-existing medical condition or taking medication that could affect taste and/or smell abilities (e.g., certain blood pressure and heart medications)
7. Allergies to foods and drinks used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Free sugar intakes | Baseline to week 12
  Percentage total energy intake (%TEI) from free sugars, measured using multiple 24-hour dietary recalls.
Adherence | week 3 to week 12
  Adherence with the dietary advice received will be assessed by self-report using online surveys.

SECONDARY OUTCOMES:
Energy intake and diet composition | Baseline to week 12
  Energy intake and nutrient composition of dietary intakes, measured using multiple 24-hour dietary recalls.
Body weight | Baseline to week 12
  Weight, in kilograms, assessed using standard digital scales.
Waist circumference | Baseline to week 12
  Waist circumference, in centimeters, measured using standard flexible tape measure.
Body fat percentage | Baseline to week 12
  Body fat percentage assessed using a bioimpedance scale.
Body mass index | Baseline to week 12
  Body mass index assessed using a standard kg/m2 measurement.
Fasted blood glucose | Baseline to week 12
  Fasted blood glucose (min 8h fast), in millimoles per litre, assessed using a prick-a-finger method and a blood glucose monitor.
Sweet food and beverage preferences | Baseline to week 12
  Preferences for sweet foods and beverages will be assessed using a taste perception test. Participants will taste commercially available several sweet and non-sweet foods and beverages and indicate how pleasant these are and how much they desire to eat these using 0-100 visual analogue scales. Higher scores indicate greater pleasantness and desire to eat.
Sweet food and beverage perceptions | Baseline to week 12
  Preferences of the sweet taste intensity will be assessed using a taste perception test. Participants will taste several commercially available sweet and non-sweet foods and beverages and indicate their sweetness intensity using 0-100 visual analogue scales. Higher scores indicate greater perceived sweetness intensity.
Sweet food and beverage choice | Baseline to week 12
  Sweet food and beverage choice will be assessed using a breakfast meal. A wide selection of commercially available sweet and non-sweet breakfast foods and beverages will be presented, with participants free to choose what and how much they consume. Sweet food and beverage choices will be measured as the weight consumed during the breakfast meal. A take-home beverage will also be offered from a selection of sweet and non-sweet beverages with the choice recorded.
Dietary advice evaluation | week 3 to week 12
  Evaluation of and perceptions of the dietary advice received will be assessed by self-report using individual questions using online surveys.
Sweet attitudes | Baseline to week 12
  Attitudes toward sugars, sweeteners, and sweet foods will be assessed using the Sweet Talk Questionnaire in six domains. The higher the score in a given domain, the more prevalent the attitude.
Self-reported quality of life | Baseline to week 12
  Physical and psychosocial functioning will be assessed using the 36-item Short Form Health Survey. Higher scores indicate greater quality of life.
Attitudes towards eating | Baseline to week 12
  General attitudes towards eating will be assessed using the Dutch Eating Behaviour Questionnaire in three domains. The higher the score in a given domain, the more prevalent the behaviour.
Dietary knowledge | Baseline to week 12
  Knowledge of dietary and sugar recommendations will be assessed via self-report using specific indvidual questions in an online questionnaire.
Adverse events | Baseline to week 12
  Adverse events will be assessed via self-report.

CONTACTS AND LOCATIONS:
Locations (1):
- Bournemouth University, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No